CLINICAL TRIAL: NCT05468775
Title: Naked Eye 3D Vision Training for the Prevention and Control of Myopia in Adolescents and Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yehong Zhuo, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021KYPJ193
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Adolescents and Children; Axial Elongation; Naked Eye 3D Vision Training; Visual Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: Naked eye 3D vision training
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Naked eye 3D vision training — 20 minutes of naked eye 3D vision training every day
  Arms: intervention group

SUMMARY:
The study used children aged 6-18 as subjects to evaluate the efficacy and safety of naked eye 3D vision training for the prevention and control of myopia in adolescents. A total of 250 subjects were recruited from Zhongshan Ophthalmology Center of Sun Yat-sen University, Shenzhen People's Hospital and Foshan Women's and Children's Hospital, with 1:1 as intervention group and control group. The study assumes that daily naked eye 3D vision training can effectively control the speed of axial elongation and the progression of myopia. The main indicators were the use of optical biometrics to detect the subjects' initial axial length and the axial length after 1 month, 3 months and 6 months of intervention. Secondary indicators were refraction, uncorrected visual acuity, best corrected visual acuity, choroidal thickness, and binocular vision.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6~18 years old (including 6 years old and 18 years old), gender is not limited;
2. Written informed consent signed by the child and legal guardian has been obtained;
3. Patients who have visited the research center in the past month, diagnosed as myopia according to the "Guidelines for the Prevention and Treatment of Myopia" issued by the General Office of the National Health Commission (Guoweiban Medical Letter [2018] No. 393), and the spherical equivalent power is -0.75 to -6.00 Diopter (D) (including -0.75 and -6.00 D);
4. Astigmatism≤4.00 D, anisometropia≤4.00 D;
5. Monocular international standard logarithmic visual acuity after spectacle correction ≥20/25;
6. The subject's guardian can understand the purpose of this study, and the subject can cooperate with the treatment and related eye examinations.

Exclusion Criteria:

1. Any eye of the subject suffers from overt strabismus, or any other pathological changes in the eyeball or acute inflammatory disease of the eye;
2. Subjects who may suffer from eye diseases that affect vision or refractive errors (such as cataract and other lens damage diseases, glaucoma, macular degeneration, keratopathy, uveitis, retinal detachment, severe vitreous opacity, etc.);
3. Systemic diseases: those with a history of immune system diseases, central nervous system diseases, Down syndrome, asthma, severe heart and lung function, severe liver and kidney dysfunction;
4. Binocular hyperopia cannot be corrected to logarithmic visual acuity of 20/25;
5. The subject has or is undergoing myopia control treatment within the past 1 month, such as atropine eye drops, orthokeratology lenses, progressive lenses, bifocal lenses, etc.;
6. Photophobia or unable to open eyes normally due to keratitis, trichiasis, trauma, etc. in any eye of the subjects;
7. Subjects participated in other clinical studies 4 weeks before enrollment;
8. For safety reasons or the interests of patients, the investigator believes that patients should not participate in other situations in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
the change of axial length | baseline, 1st months, 3rd months, 6th months
  mm

SECONDARY OUTCOMES:
the change of vision | baseline, 1st months, 3rd months, 6th months
  Diopter
the change of choroidal thickness | baseline, 1st months, 3rd months, 6th months
  mm
the change of adjustment range | baseline, 1st months, 3rd months, 6th months
  Diopter
the change of adjust sensitivity | baseline, 1st months, 3rd months, 6th months
  cycle per minute

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie R, Zhao F, Yu J, Luo B, Jiang Z, Qiu X, Cao Y, Yang Y, Chen K, Zhang Y, Luo X, Wang Z, Zhu Y, Zhuo Y. Naked-Eye 3-Dimensional Vision Training for Myopia Control: A Randomized Clinical Trial. JAMA Pediatr. 2024 Jun 1;178(6):533-539. doi: 10.1001/jamapediatrics.2024.0578. PMID 38587852